CLINICAL TRIAL: NCT01536210
Title: Randomized, Double-Blind, Placebo-control, Multicenter Study, the Efficacy and Safety of Combination of Ginkgo Extract and Ginseng Extract(YY-162)in Children With ADHD(Attention Deficit Hyperactivity Disorder)in 8 Weeks
Brief Title: Efficacy and Safety Study of Combination of Ginkgo Extract and Ginseng Extract in Children With ADHD(Attention Deficit Hyperactivity Disorder)
Acronym: ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YY-162 (b)
Record Dates: First submitted 2012-01-09; First posted 2012-02-20 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Mental Disorders
Keywords: ADHD(attention Deficit Hyperactivity Disorder)
MeSH Terms: conditions — Mental Disorders; Attention Deficit Disorder with Hyperactivity | interventions — YY162; Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YY-162 (Experimental): YY-162(Ginkgo Extract 30mg + Ginseng Extract 50mg)
  1T/Three times a day(Tid) for 8 weeks, PO medication
  Interventions: Drug: YY-162
- Placebo (Placebo Comparator): Placebo 1T /Three times a day(Tid) for 8 weeks, PO medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YY-162 — YY-162(Ginkgo extract 30mg + Ginseng extract 50mg) 1T/Three times a day(Tid) for 8 weeks, PO medication
  Other Names: combination of Ginkgo extract and Ginseng extract
  Arms: YY-162
Drug: Placebo — Placebo 1T/ Three times a day (tid) for 8 weeks, PO medication
  Arms: Placebo

SUMMARY:
This study will evaluate clinical efficacy and safety of treatment with YY-162 in children with ADHD.

DETAILED DESCRIPTION:
This is Double-Blind, two arms, multi-center, Interventional, 8 weeks study starting with YY-162(Combination of Ginkgo extract and Ginseng extract)in children with ADHD. Assessment of efficacy and safety will be performed at the baseline, weeks 2, 4 and 8. At the first visit, a full psychiatric history, demographic date and physical examination will be undertaken. Throughout the study, the following procedures, documentations and evaluations will performed; K-ARS, IOWA conner's rating scale, CGI-S/I, ATA, Children's color trails test and stroop test, intelligence test(from KEDI-WISC)and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Mele and female subjects aged from 6 to 15
* Subjects must meet DSM-IV criteria for ADHD based-on the K-Schedule for affective disorder and schizophrenia(K-SADS-PL-K)interview
* Subjects signed a written consent form voluntarily
* Patient's assent to participate in the study and written informed consent form signed by one of the parents, parent surrogates or legal guardian.
* Subjects who can keep visit schedule and whose parent/parent surrogates or legal guardian can willingly complete assessments defined in the study protocol.
* Subjects/parents, parent surrogates or legal guardian who can understand the participation of the study and voluntarily withdraw from the study at any time.

Exclusion Criteria:

* Subjects who have difficulty swallowing tablet.
* Subjects who have known allergy to plant extracts.
* Subjects who meet DSM-IV diagnostic criteria for current major depressive disorder or anxiety disorder requiring drug therapy.
* Subjects who have any history of bipolar disorder, psychotic disorder, and substance use disorder, have been diagnosed with a pervasive developmental disorder, organic brain disease and seizure disorder.
* Subjects who have significant suicidal ideation.
* Subjects with mental retardation.
* Subjects with Tourette's syndrome requiring drug therapy.
* Subjects who have been administrated Methylphenidate or Atomoxetine within recent 3 months and Ginkgo extract or Ginseng extract within recent 1 month.
* Subjects who currently have a significant medical conditions(e.g. diseases of cardiovascular, hepatic, renal, respiratory, glaucoma)
* Subjects who have abnormalities in the ECG or show clinically significant abnormalities of laboratory results including serum chemistries and hematology.
* subjects who are currently taking alpha-2 adrenergic receptor agonist, antidepressant, antipsychotic, benzodiazepines, modafinil, anticonvulsant.
* subjects who receive psychosocial treatment during the drug trial.
* Subjects who are not able to swallow the study drug.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Korea-ADHD Rating scale | within the first 8 weeks (plus or minus 5 days) after adminitration
  Validated questionnaire about core ADHD symptoms(Korea-ADHD Rating scale) filled out by patents at baseline, after 8 weeks.

SECONDARY OUTCOMES:
IOWA conner's rating scale | baseline, after 2, 4, and 8 weeks
  Validated questionnaire about core ADHD symptoms(IOWA Conner's rating scale) filled out by parents at baseline, after 2,4 weeks and closeout
Clinical Global Impression(Severity and Improvement) | baseline, after 2, 4, and 8 weeks
  Clinical Global Impression(Severity and Improvement)rated by treating physician at baseline, after2,4 weeks and closeout
Advanced Test of Attention | baseline and 8 weeks
  Advanced Test of Attention and baseline and closeout Attention Diagnostic system(visual and auditory) at baseline and closeout
children's color trails test and stroop test | baseline and 8 weeks
  Children's color trails test and stroop test at baseline and closeout
Intelligence test(from KEDI-WISC) | screening and 8 weeks
  Intelligence test(from KEDI-WISC)at screening and closeout

CONTACTS AND LOCATIONS:
Overall Officials: SooChurl Cho, MD, PhD, Principal Investigator — Seoul National University Hospital; HyunJu Hong, MD, PhD, Principal Investigator — Hallym University Hospital; EunJin Park, MD, Principal Investigator — Inje University
Locations (3):
- South Korea (3):
  - Hallym University Hospital, Anyang-si
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Result] Lyon MR, Cline JC, Totosy de Zepetnek J, Shan JJ, Pang P, Benishin C. Effect of the herbal extract combination Panax quinquefolium and Ginkgo biloba on attention-deficit hyperactivity disorder: a pilot study. J Psychiatry Neurosci. 2001 May;26(3):221-8. PMID 11394191
- See also: Effect of the herbal extract combination Panax quinquifolius and Ginkgo biloba on attention-deficit hyperactivity disorder: a pilot study — http://www.ncbi.nlm.nih.gov/pubmed